

# Non-Interventional Study Protocol B3461058

# Prevalence and characteristics of transthyretin amyloidosis in patients with left ventricular hypertrophy of unknown etiology TTRACK

Statistical Analysis Plan (SAP)

Version: 2

Author: PPI

**Date**: 06-Jul-2022

# TABLE OF CONTENTS

| A | BBREVIATIONS | 4 |
|---|---|---|
| 1 | AMENDMENTS FROM PREVIOUS VERSION(S) | 5 |
| 2 | INTRODUCTION | 5 |
| | 2.1 STUDY DESIGN | SECONT S |
| | 2.2 STUDY OBJECTIVES | 7 |
| 3 | INTERIM ANALYSES | 8 |
| 4 | HYPOTHESES AND DECISION RULES | 8 |
| | 4.1 STATISTICAL HYPOTHESES | |
| 5 | ANALYSIS SETS/POPULATIONS | 9 |
| | 5.1 FULL ANALYSIS SET Full Analysis Set 1 – Primary population Full Analysis Set 2 – All FAS1 patients with positive scintigraphy (grade 1, 2 or 3 Full Analysis Set 3 – All FAS2 patients with positive scintigraphy grade 2 or 3 (Cardiac amyloidosis) 5.2 SAFETY ANALYSIS SET 5.3 SUBGROUPS | 9<br>3) 9<br>9<br>9 |
| 6 | ENDPOINTS AND COVARIATES | . 10 |
| | 6.1 EFFICACY/EFFECTIVENESS ENDPOINTS. 6.2 SAFETY ENDPOINTS. 6.3 OTHER ENDPOINTS. Primary endpoint. Secondary endpoints. 6.4 COVARIATES. | . 10<br>. 10<br>. 10<br>. 10 |
| 7 | HANDLING OF MISSING VALUES | . 13 |
| 8 | STATISTICAL METHODOLOGY AND STATISTICAL ANALYSES | . 13 |
| | 8.1 STATISTICAL METHODS 8.2 STATISTICAL ANALYSES Safety analyses Analysis of primary and secondary objectives Other analyses | . 14<br>. <i>14</i><br>. <i>14</i> |
| 9 | | |
| | PFIZER CONFIDENTIAL | |

| 10 | REFERENCES. 2 | 22 |
|----|-----------------------------------------|----|
| | APPENDICES 2 | |
| | 1.1 Appendix 1: Data Derivation Details | |

# **ABBREVIATIONS**

| Abbreviation | Definition |
|---|---|
| <sup>99</sup> mTc-DPD | 99mTechnetium-3,3-diphosphono-1,2-propanodi-carboxylic acid |
| <sup>99</sup> mTc-PYP | 99mTechnetium-pyrophosphate |
| <sup>99</sup> mTc-HMDP | 99mTechnetium-hydroxymethylene diphosphonate |
| AA | Serum Amyloid A Protein |
| AE | Adverse event |
| AICD | Automatic Implantable Cardiac Defibrillator |
| AL | Light chain amyloidosis |
| ATTR | Transthyretin amyloidosis |
| ATTR-CM | Transthyretin amyloid cardiomyopathy |
| ATTRv | Variant transthyretin related amyloidosis |
| ATTRwt | Wild type transthyretin related amyloidosis |
| AVA | Aortic valve area |
| CI | Confidence interval |
| CM | Cardiomyopathy |
| CTS | Carpal Tunnel syndrome |
| ECG | Electrocardiogram |
| ЕСНО | Echocardiography |
| e-CRF | Electronic Case Report Form |
| FAS | Full analysis set |
| HCM | Hypertrophic cardiomyopathy |
| IQR | Interquartile Range |
| LGE | Late gadolinium enhancement |
| LV | Left ventricular |
| LVH | Left ventricular hypertrophy |
| LVOTO | Left ventricular outflow tract obstruction |
| MRI | Magnetic resonance imaging |
| MWT | Maximal wall thickness |
| NI | Non-interventional |
| NT-proBNP | N-terminal pro-brain natriuretic peptide |
| PN | Polyneuropathy |
| PT | Preferred term |
| SAE | Serious adverse event |
| SAF | Safety analysis set |
| SCD | Sudden cardiac death |
| sFLC | Serum Free Light Chain |
| SOC | System Organ Class |
| SPECT | Single Photon Emission Computed Tomography |
| TTR | Transthyretin |

## 1 AMENDMENTS FROM PREVIOUS VERSION(S)

| Version | Effective Date | Change Type<br>(New, Revise,<br>Admin) | Summary of Revisions |
|---|---|---|---|
| 1 | 27-Apr-2020 | New | |
| 2 | 06-Jul-2022 | Revise | <ul> <li>Wording modified in line with clarifications in protocol amendment 2</li> <li>To add sensitivity analyses to assess the impact of: <ul> <li>using a SPECT</li> <li>no longer using a centralized lab</li> </ul> </li> <li>Subgroups analyses added</li> <li>To add scintigraphy discrepancies analysis</li> </ul> |

#### 2 INTRODUCTION

Note: in this document any text taken directly from the non-interventional (NI) study protocol is *italicised*.

The main purpose of this study is to determine the prevalence of transthyretin amyloid cardiomyopathy (ATTR-CM) among patients admitted due to left ventricular hypertrophy (LVH) of unknown etiology when radionuclide bone scintigraphy or single photon emission computed tomography (SPECT) is used.



Figure 1. Diagnostic algorithm for patients with suspected amyloid cardiomyopathy (Gillmore 2016).

#### 2.1 STUDY DESIGN

TTRACK is an epidemiological multicenter and multinational study.

#### **Study population**

This study will include patients with LVH from undiagnosed etiology and the following inclusion/exclusion criteria:

#### 1. Inclusion criteria:

- a. Patient signed inform consent.
- b. Males and Females.
- c.  $Age \ge 50$  years.
- d. Left ventricular hypertrophy (LVH) defined as end-diastolic LV maximum wall thickness (MWT)  $\geq$ 15mm in Echocardiogram.

e. Plan to undergo or recently underwent radionuclide bone scintigraphy and/or SPECT with any of the following radio labelled tracers: 99mTc-DPD or 99mTc-

PYP or <sup>99m</sup>Tc-HMDP.

Scintigraphy will be defined at each site according to the standard grading:

Grade 0 = absent cardiac uptake

 $Grade\ 1 = mild\ uptake\ less\ than\ bone$ 

 $Grade\ 2 = moderate\ uptake\ equal\ to\ bone$ 

 $Grade\ 3 = high\ uptake\ greater\ than\ bone$ 

#### 2. Exclusion criteria

a. Etiological diagnosis explaining the LVH prior to patient inclusion (eg, Sarcomeric HCM, Myeloma, Fabry disease, Sarcoidosis, any type of amyloidosis [AA, AL, TTR\*\*])

\*\* TTR diagnosis at exclusion criteria: Direct relative (siblings or parents) of a carrier with a known hereditary mutation in the TTR gene or any patient already diagnosed by any of the following: cardiac fixation at the bone scintigraphy, TR mutation at the genetic testing, biopsy with amyloidosis (positive red congo) and positive TTR staining.

b. Severe aortic stenosis defined as aortic valve area (AVA) < 1.0 cm<sup>2</sup>

#### Data source

Data will come from medical records and will be collected in routine clinical practice. As an epidemiological study, there are no specific requirements with regard to patient procedures to be performed or the treatment regimen. Data from each patient will be reported on an electronic case report form (e-CRF).

#### **Treatment/cohort labels**

NA

# 2.2 STUDY OBJECTIVES

#### 1. Primary objective

• To assess the prevalence of patients with cardiac fixation at the radionuclide bone scintigraphy and/or Single Photon Emission Computed Tomography (SPECT) performed with 99mTc-DPD or 99mTc-PYP or 99mTc-HMDP\* among patients with (left ventricular hypertrophy) LVH from undiagnosed etiology;

## 2. Secondary objectives

• To assess the prevalence of Light Chain Amyloidosis (AL) or Transthyretin amyloid (ATTR) amyloidosis in patients with cardiac fixation at the bone scintigraphy (visual grade 1 to 3) and/or SPECT;

- To assess the prevalence of hereditary (ATTRv) and wild-type (ATTRwt) ATTR amyloidosis in patients diagnosed with ATTR amyloidosis;
- To describe TTR genetic mutations\*\* in patients with ATTRv amyloidosis;
- To assess the prevalence of patients with familial history of known cardiomyopathy (CM), polyneuropathy (PN), sudden cardiac death (SCD) among their relatives (ie, parents, siblings and  $2^{nd}/3^{rd}$  degree grade family members);
- To assess the prevalence in patients with cardiac fixation at the bone scintigraphy or SPECT of concomitant signs or symptoms of ATTR amyloidosis, ie,:
  - Sensori-motor Polyneuropathy (PN);
  - Carpal Tunnel syndrome (CTS);
  - o Autonomic dysfunction;
  - Cardiological manifestations;
  - o Laboratory signs;
- To compare the clinical and biochemical characteristics between patients with positive scintigraphy (cardiac fixation at the bone scintigraphy grade 1, 2 or 3) and/or SPECT;
- To assess the level of discrepancy in the evaluation of the scintigraphy and/or SPECT images by different evaluators.
- \* Bisphosphonate (99mTc-DPD/99mTc-PYP/99mTc-HMDP) Scintigraphy
- \*\* Variant and pathogenic mutation by sequencing the coding parts

#### 3 INTERIM ANALYSES

An interim analysis of the data collected was planned for all the variables as soon as 75 patients will be selected with a scintigraphy grade 1, 2 or 3 and with completed e-CRF. This interim analysis was finally not performed.

In addition, an interim analysis was performed for publication purpose, all patients screened until the May 11<sup>th</sup> 2020 were included in this analysis. Considering the expected number of patients with a scintigraphy grade 1, 2 or 3, all analyses described in this SAP were done, except multivariate analyses planned in 0.

#### 4 HYPOTHESES AND DECISION RULES

#### 4.1 STATISTICAL HYPOTHESES

TTRACK is a non-interventional and uncontrolled study. In that sense, there is no inferential hypothesis that will serve for a claim.

#### 4.2 STATISTICAL DECISION RULES

The analysis of this study will be mainly descriptive. However, factors associated to ATTR will be identified using a multivariate analysis. All statistical tests will be exploratory in nature.

#### 5 ANALYSIS SETS/POPULATIONS

#### 5.1 FULL ANALYSIS SET

#### <u>Full Analysis Set 1 – Primary population</u>

Full Analysis Set 1 (FAS1) includes all patients who meet eligibility (inclusion/exclusion) criteria and with a radionuclide bone scintigraphy and/or SPECT performed with 99mTc-DPD/99mTc-PYP/99mTc-HMDP.

# Full Analysis Set 2 – All FAS1 patients with positive scintigraphy (grade 1, 2 or 3)

Full Analysis Set 2 (FAS2) is a subset of FAS1 patients with grading of cardiac retention equal to grade 1, grade 2 or grade 3.

Analysis of group 1 vs group 2&3 independently and grouped will be performed Patients with grade 1 will be considered od "undetermined etiology"

# <u>Full Analysis Set 3 – All FAS2 patients with positive scintigraphy grade 2 or 3 (Cardiac amyloidosis)</u>

Full Analysis Set 3 (FAS3) is a subset of FAS2 patients with grading of cardiac retention equal to grade 2 or grade 3.

**FAS 3.1** Patients with grade 2-3 **without** monoclonal protein abnormalities (ATTR amyloidosis)

**FAS 3.2** Patients with grade 2-3 **with** monoclonal protein abnormalities (Undefined etiology, cardiac ATTR amyloidosis, or MGUS or AL Amyloidosis). Monoclonal protein abnormalities if defined as Positive IFE (serum and/or urine) or positive FLC (See definition in section 6.3).

#### 5.2 SAFETY ANALYSIS SET

Safety Analysis Set (SAF) includes all enrolled patients.

#### 5.3 SUBGROUPS

Some secondary endpoints (See table in section 8.2) will also be described by the following subgroup:

• ATTRv: ATTR patients with a ATTR gene sequencing with variant transthyretin will be considered as ATTRv.

ATTRwt: ATTR patients with a ATTR gene sequencing with a result of « No

Mutation » will be considered as ATTRwt

#### 6 ENDPOINTS AND COVARIATES

#### 6.1 EFFICACY/EFFECTIVENESS ENDPOINTS

NA

#### 6.2 SAFETY ENDPOINTS

Adverse events (AE) will be coded using MedDRA version 20.0 or later.

#### 6.3 OTHER ENDPOINTS

#### Primary endpoint

Patients with cardiac fixation at the radionuclide bone scintigraphy and/or SPECT performed with 99mTc-DPD or 99mTc-PYP or 99mTc-HMDP will be defined as patients with a cardiac retention of grade 1, grade 2 or grade 3.

Patients without cardiac fixation at the radionuclide bone scintigraphy performed and/or SPECT with 99mTc-DPD or 99mTc-PYP or 99mTc-HMDP will be defined as patients with a cardiac retention of grade 0.

#### **Secondary endpoints**

- 1. Presence of Transthyretin amyloid (ATTR) or patients with suspicion of MGUS / Light Chain Amyloidosis (AL)
- Patients with grade 2 or 3 at scintigraphy will be considered "Cardiac amyloidosis patients"
  - Patients with grade 2 or 3 at scintigraphy without monoclonal protein abnormalities will be considered patients with **ATTR amyloidosis**
  - Patients with grade 2 or 3 at scintigraphy with monoclonal protein abnormalities
    will be considered of the population of patients with suspicion of MGUS or AL
    amyloidosis
- Patients with grade 1 at scintigraphy will be considered as "undetermined"

Monoclonal protein abnormalities are defined as patients with positive IFE (Immunofixation electrophoresis) (serum and urine) or with abnormal FLC (free light chain) ratio:

| | eGFR | | | |
|--------------------|-------------------------|-------|-------|-------|
| | >60 45-<60 30-<45 <30 | | | |
| Abnormal FLC ratio | ≥1.65 | ≥1.92 | ≥2.06 | ≥2.17 |
| Normal FLC ratio | <1.65 <1.92 <2.06 <2.17 | | | |

# eGFR will be calculated with MDRD formula:

 $\overline{\text{GFR (mL/min/1.73 m}^2)} = 175 \times (\overline{\text{Serum }}_{\text{creatinine}})^{-1.154} \times (\overline{\text{Age}})^{-0.203} \times (0.742 \text{ if female}) \times (1.212 \text{ if African American) (conventional units)}$ 

# 2. Presence of hereditary (ATTRv) and wild-type (ATTRwt) ATTR

ATTR patients with a ATTR gene sequencing with variant transthyretin will be considered as ATTRv.

ATTR patients with a ATTR gene sequencing with a result of « No Mutation » will be considered as ATTRwt.

# 3. Presence of familial history of known cardiomyopathy (CM), polyneuropathy (PN), sudden cardiac death (SCD)

Family history for each disease will be considered for  $1^{st}$  degree parent, siblings and  $2^{nd}/3^{rd}$  grade family.

# 4. Senso-motor Polyneuropathy

Patients with at least one red flag in the neurological part of the ATTR-Amyloidosis red flags e-CRF part will be considered as patients with a senso-motor Polyneuropathy.

#### 5. Carpal Tunnel syndrome (CTS)

Patients with a CTS will be patients with a bilateral or unilateral CTS. Patients without CTS will be patients with a "NO" to the question "Carpal tunnel syndrome symptoms"

#### 6. Autonomic dysfunction

Patients with autonomic dysfunction will be patients with at least one autonomic sign or autonomic symptom = "Yes"

# 7. Cardiological manifestations

Patients with cardiological signs will be defined as patients with at least one of the following criteria fulfilled:

| Criterion | Value |
|---|---|
| In Cardiological assessments part of the e-CRF | |
| Atrial Fibrillation | Yes permanent |
| Pacemaker | Yes |
| AICD | Yes |
| In MRI part of the e-CRF | |
| LGE | Positive |
| In ECG part of the e-CRF | |
| Sinus rhythm | No |
| PR interval | < 80 ms or > 350 ms |
| QRS interval | < 60 ms or > 250 ms |
| Sokolow index | < 1 mm or > 70 mm |
| Pseudo-MI pattern | Yes |
| PPOr precordial R wave progression | Yes |
| LBBB | Ticked |
| RBBB | Ticked |
| Paced | Ticked |
| Intraventricular conduct delay | Ticked |
| LVOT | Yes |
| If longitudinal strain is done, strain apical preserved | Yes |
| LV end-diastolic diameter | < 20 mm or > 80 mm |
| MWT | < 15 mm or > 100 mm |
| MWT at septum | < 3 mm or > 50 mm |
| MWT posterior wall | < 3 mm or > 50 mm |
| LV mass index | $< 40 \text{ g/m}^2 \text{ or} > 160 \text{ g/m}^2$ |
| Maximal aortic velocity | > 5 m/s |
| Mean gradient of Aortic valvular stenosis | > 70 mmHg |
| Area of Aortic valvular stenosis | $< 0.2 \text{ cm}^2 \text{ or} > 3 \text{ cm}^2$ |

#### 8. Laboratory signs

Patients with at least one blood test laboratory result out of range will be considered as patients with laboratory signs.

- For creatinine, patients with a value lower than 45  $\mu$ mol/L or higher than 104  $\mu$ mol/L will be considered as out of range
- For haemoglobin, patients with a value lower than 11,5 g/dL or higher than 16. g/dL will be considered as out of range
- For BNP, patients with a value higher than 100 pg/mL will be considered as out of range
- For NTproBNP, patients with a higher than 125 pg/mL will be considered as out of range
- For Troponin I, patients with a value higher than 26 pg/mL will be considered as out of range

out of range

- For Troponin T, patients with a value higher than 14 pg/mL will be considered as

#### 9. Coexistence of typical neurological signs / symptoms

Patients with only one redflag / patients with two redflags / patients with at least three redflags.

#### 6.4 COVARIATES

- Grade (0, 1, 2, 3) and for grade 2&3 pooled together
- Age in class  $50 \le 60$ ;  $> 60 \le 70$  years;  $> 70 \le 80$  years; > 80 years]
- Gender (Male/Female)
- Cardiological symptomatology (Yes/No, where patient with a cardialogical symptomatology are defined as patient with a least one cardiological manifestation (point 7 in 0)
- High Creatinine, high BNP and high NTproBNP (See Section 6.3, § 8)

#### 7 HANDLING OF MISSING VALUES

Missing data will not be imputed.

# 8 STATISTICAL METHODOLOGY AND STATISTICAL ANALYSES8.1 STATISTICAL METHODS

Quantitative variables will be described using number of filled and missing data, mean, standard deviation, median, 1<sup>st</sup> and 3<sup>rd</sup> quartiles, minimum and maximum. The 95%CI of the mean will also be provided, assuming a normal distribution. In case of departure from normality, results will be interpreted based on median and Interquartile Range (IQR).

Qualitative variables will be described using number of filled and missing data and, for each modality, the frequency and percentage (referring to filled data). A 95% confidence interval (CI) will be associated to binomial proportions using the Wilson score method.

Factors associated to an outcome of interest (ATTR vs other and ATTRwt vs ATTRv within patients diagnosed with ATTR-CM) will be identified using univariate logistic regression models. A separate logistic regression model will be created for each factor (as well as covariates described in section 6.4). If the variable is significantly associated to the outcome at the 10% level then the factor will be put forward into a multivariate model. Once the univariate model selection is complete, backwards selection will be used to remove factors from the multivariate model which do not have a significant p value at the 5% level. The covariate with the highest p value will be removed in turn until all factors have a p value less than 0.05. If a significant interaction is found then the individual factors of this interaction will be kept in the model, regardless of their p value. A significant interaction is tested for between all variables in the multivariate model.

Furthermore, a table showing all of the 95% confidence intervals and p values for the odds ratios coming from the univariate and multivariate models will be created.

#### 8.2 STATISTICAL ANALYSES

Analyses will be provided overall and by subgroup defined in section 5.3.

#### **Safety analyses**

The safety analysis will be performed on the SAF population. AEs will be listed based on data recorded in the eCRF. A flag will be added to the AEs listing to identify patients who meet eligibility (inclusion/exclusion) criteria and with a radionuclide bone scintigraphy and/or SPECT performed with99mTc-DPD/99mTc-PYP/99mTc-HMDP. No statistical test will be performed.

## Analysis of primary and secondary objectives

For each objective, a percentage/prevalence with its 95%CI will be assessed overall and in the sub-groups defined in section 5.3 if pertinent.

| Endpoints | Population or |
|---|---|
| | Subgroup |
| Percentage of patients with cardiac fixation at the radionuclide | FAS1 |
| bone scintigraphy and/or SPECT performed with 99mTc-DPD or | |
| 99mTc-PYP or 99mTc-HMDP among patients with (left ventricular | |
| hypertrophy) LVH from an undiagnosed etiology | |
| Prevalence of Transthyretin amyloid (ATTR) or patients with | FAS1 |
| suspicion of MGUS / AL amyloidosis | |
| Prevalence of hereditary (ATTRv) and wild-type (ATTRwt) | FAS2 & 3 |
| ATTR amyloidosis in patients with positive scintigraphy | (including 3.1 |
| | and 3.2) |
| Prevalence of TTR genetic mutation in patients with positive | FAS2 & 3 |
| scintigraphy | (including 3.1 |
| | and 3.2) |
| Prevalence of patients with familial history of known | FAS1, 2 & 3 |
| cardiomyopathy (CM), polyneuropathy (PN), sudden cardiac | (including 3.1, |
| death (SCD) among their relatives (parents, siblings and 2 <sup>nd</sup> /3 <sup>rd</sup> | 3.1(ATTRv), |
| grade family) | 3.1(ATTRwt) |
| | and 3.2) |
| Prevalence of patients with Senso-motor Polyneuropathy | FAS2 & 3 |
| | (including 3.1, |
| | 3.1(ATTRv), |
| | 3.1(ATTRwt) |
| | and 3.2) |

| Endpoints | Population or<br>Subgroup |
|---|---|
| Prevalence of patients with CTS | FAS2 & 3<br>(including 3.1,<br>3.1(ATTRv),<br>3.1(ATTRwt)<br>and 3.2) |
| Prevalence of patients with autonomic dysfunction | FAS2 & 3<br>(including 3.1,<br>3.1(ATTRv),<br>3.1(ATTRwt)<br>and 3.2) |
| Prevalence of patients with cardiological manifestations | FAS2 & 3<br>(including 3.1,<br>3.1(ATTRv),<br>3.1(ATTRwt)<br>and 3.2) |
| Prevalence of patients with laboratory signs | FAS2 & 3<br>(including 3.1,<br>3.1(ATTRv),<br>3.1(ATTRwt)<br>and 3.2) |
| Description of the clinical and biochemical characteristics between patients with positive scintigraphy (cardiac fixation at the bone scintigraphy grade 1, 2 or 3) and/or SPECT (See section 0 § 3). | FAS2 & 3<br>(including 3.1,<br>3.1(ATTRv),<br>3.1(ATTRwt)<br>and 3.2) |
| Discrepancy in the evaluation of the scintigraphy and/or SPECT images by different evaluators (See section 0 § 7) | FAS1 |

# **Other analyses**

# 1. Patient characteristics

A full description of patient characteritics will be provided in the FAS1.

**2.** <u>Analysis of redflags</u>
The prevalence of each redflag will be assessed in the FAS 1, 2 & 3 population.

#### 3. Description of variables of interest

Variables of interest are all variables collected in the CRF (including Kappa, Lambda, IgG, IgA and IgM rates from monoclonal protein studies).

- Variables of interest will be described in the FAS2 & 3 population in patients with 1, 2 or 3 redflags.
- Variables of interest will be described in the FAS1 population in patients with grade 0/1/2/3.
- Variables of interest will be described in the FAS2 & 3 population in patients with ATTRv and ATTRwt.

# 4. <u>Comparaison between patients with final diagnosis of ATTR-CM and screened patients</u>

Patients with a final diagnosis of ATTR-CM will be compared with the other "negative" screened patients in order to highlight possible diagnostic TTR-Amyolosis red flags

## 5. Factors associated to positive scintigraphy

Factors associated to positive scintigraphy will be identified in the FAS1 by univariate and multivariate logistic regression. This analysis will be performed in the FAS1 population and will include all variables collected in the CRF for both positive and negative scintigraphy. Clinical laboratories will be excluded from this analysis as only available for positive scintigraphy.

#### 6. Factors associated to grade 2-3 scintigraphy and ATTR-CM

Factors associated to grade 2 or 3 will be identified in the FAS1 by univariate and multivariate logistic regression (compared with negative patients). This analysis will be performed in the FAS1 population and will include all variables collected in the CRF for both positive and negative scintigraphy. Clinical laboratories will be excluded from this analysis as only available for positive scintigraphy. The same analysis will be repeated to identify factors associated to ATTR-CM (FAS 2 & 3).

#### 7. Scintigraphy discrepancies analysis

Discrepancy in the evaluation of the scintigraphy and/or SPECT images by different evaluators will be analyzed as follow:

• Between site and 1st evaluator:

Cross tabulation between the two evaluators

| Scintigraphy or SPECT images | tigraphy or SPECT images Site evaluation | | | | |
|---|---|---|---|---|---|
| 1 <sup>st</sup> external evaluator | Grade | 0 | 1 | 2 | 3 |
| | 0 | | | | |
| | 1 | | | | |
| | 2 | | | | |
| | 3 | | | | |

All percentages of discrepancies will be provided. A weighted Kappa coefficient (measure of interrater agreement) will be provided with 95% confidence limits and exact test for the kappa coefficient.

- Between 1<sup>st</sup> and 2<sup>nd</sup> evaluators (in case there is a discrepancy between site evaluation and 1<sup>st</sup> external evaluator), same analyses will be performed.
- A listing of all individual patients will be provided for all discrepancies (site and the 2 external evaluations).

#### 8. Sensitivity analyses

- 1) Impact of protocol amendment 2 Use of SPECT
  The prevalence of patients with cardiac fixation at the radionuclide bone scintigraphy and/or Single Photon Emission Computed Tomography (SPECT) performed with 99mTc-DPD or 99mTc-PYP or 99mTc-HMDP\* among patients with (left ventricular hypertrophy) LVH from undiagnosed etiology will be calculated in patients included before protocol amendement and in patients included after protocol amendement (Amendement 2 Date: 11-Feb-2020). The percentage and its 95% CI will be provided.
- 2) Impact of protocol amendment 2 No longer using a centralized lab

  The prevalence of patients with laboratory signs will be calculated in patients included before protocol amendement and in patients included after protocol amendement (Amendement 2 Date: 11-Feb-2020). The percentage and its 95% CI will be provided.

## 9 LIST OF TABLES AND TABLE SHELLS

A list of tables will be provided in a separate document. An example of some table shells is presented below:

Table 15.1.1 Number and Percentage of Patients in Each Analysis Set

| Analysis | | Grade 0 | Grade 1 | Grade 2 | Grade 3 | Unknown grade | Total |
|---|---|---|---|---|---|---|---|
| Set | | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Selected | No | | | | | | xx (xx.x%) |
| | Yes | | | | | | xx (xx.x%) |
| FAS1 | No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Yes | | | | | xx (xx.x%) | xx (xx.x%) |
| FAS2 | No | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Yes | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| FAS3 | No | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Yes | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| FAS4 | No | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Yes | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Safety Set | No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Yes | xx (xx.x%) | | | | xx (xx.x%) | xx (xx.x%) |

. . .

Table 15.1.2 Demography and Baseline Characteristics – FAS1, 2

| | | | | FA | S 2 | | |
|---|---|---|---|---|---|---|---|
| Variables | | Grade 0 | Grade 1 | Grade 2 | Grade 3 | Grade 1 or 2<br>or 3 | Total (FAS 1) |
| | | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | |
| Age (years) | N | xx | xx | xx | xx | xx | xx |
| | Mean ± SD | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ |
| | Median | xx.x | XX.X | xx.x | XX.X | xx.x | xx.x |
| | Q1; Q3 | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x |
| | Min. ; Max. | xx;xx | xx;xx | xx;xx | XX;XX | xx;xx | xx;xx |
| | Missing | X | х | х | X | X | х |
| Age (in class) | [50 - 55]<br>years | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | ]55 - 60]<br>years | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | ]60 - 65]<br>years | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | ]65 - 70]<br>years | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | ]70 - 75]<br>years | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | PFIZ | ZER CONFIDE | ENTIAL | | | |

| | ]75 - 80]<br>years | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
|---|---|---|---|---|---|---|---|
| | over 80 years | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Gender | Missing | xx | xx | xx | xx | xx | xx |
| | Male | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| | Female | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Weight (kg) | N | xx | xx | xx | xx | xx | XX |
| | Mean ± SD | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | xx.x ± x.x |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Q1; Q3 | XX.X; XX.X | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x | XX.X;XX.X |
| | Min. ; Max. | XX;XX | xx;xx | xx;xx | xx;xx | xx;xx | xx ; xx |
| | Missing | X | x | x | x | x | Х |
| BMI (kg/m²) | N | xx | xx | xx | xx | xx | XX |
| | Mean ± SD | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ | xx.x ± x.x |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Q1 ; Q3 | XX.X; XX.X | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x | XX.X ; XX.X |
| | Min. ; Max. | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx |

Table 15.1.2 Demography and Baseline Characteristics – FAS 2&3

| | | FAS 3 | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Variables | | Grade 1 | ATTRwt | ATTRv | ATTR<br>(=FAS 3.1) | FAS 3.2 | All FAS 3 | Total (=FAS |
| | | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | |
| Age<br>(years) | N | xx | xx | xx | xx | xx | xx | xx |
| | Mean ±<br>SD | xx.x ± x.x | xx.x ± x.x | XX.X ± X.X | xx.x ± x.x | XX.X ± X.X | xx.x ± x.x | xx.x ± x.x |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Q1; Q3 | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x | xx.x; xx.x |
| | Min. ;<br>Max. | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx |
| | Missing | x | x | x | X | x | х | Х |
| Age (in class) | [50 - 55]<br>years<br>]55 - 60]<br>years | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | ]60 - 65]<br>years | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | | PFIZEI | R CONFIDE | NTIAL | | | |

| | ]65 - 70]<br>years | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
|---|---|---|---|---|---|---|---|---|
| | ]70 - 75]<br>years | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | ]75 - 80]<br>years | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | over 80<br>years | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Gender | Missing | XX | XX | XX | XX | XX | XX | xx |
| | Male | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Female | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Weight | N | XX | XX | XX | XX | XX | XX | XX |
| (kg) | Mean ±<br>SD | xx.x ± x.x | xx.x ± x.x | xx.x ± x.x | xx.x ± x.x | xx.x ± x.x | xx.x ± x.x | xx.x ± x.x |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Q1 ; Q3 | xx.x; xx.x | XX.X; XX.X | XX.X; XX.X | xx.x; xx.x | XX.X; XX.X | xx.x; xx.x | xx.x; xx.x |
| | Min. ;<br>Max. | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx |
| | Missing | x | x | x | x | x | x | x |
| BMI | N | XX | XX | XX | XX | XX | xx | XX |
| (kg/m²) | Mean ±<br>SD | xx.x ± x.x | xx.x ± x.x | xx.x ± x.x | xx.x ± x.x | xx.x ± x.x | xx.x ± x.x | xx.x ± x.x |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Q1 ; Q3 | xx.x; xx.x | XX.X; XX.X | XX.X;XX.X | xx.x; xx.x | XX.X;XX.X | xx.x; xx.x | xx.x;xx.x |
| | Min. ;<br>Max. | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx | xx ; xx |
| | Missing | х | х | Х | Х | Х | x | x |

. . .

Table 15.2.1 Prevalence of Patients with Cardiac Fixation at the Radionuclide Bone Scintigraphy and / or SPECT Performed – FAS1

| Variable(s) | Total<br>(N=XX) |
|---|---|
| Prevalence of patients with cardiac fixation at the radionuclide bone scintigraphy and /or SPECT performed | xx (xx.x%) |
| IC95% | [xx.x% - xx.x%] |

...

Table 15.2.2 Factors Associated to Positive Scintigraphy (Logistic Regression Model) – FAS1

| | Positive S | cintigraphy | Univariate Analysis | | Multivariate Analysis | |
|---|---|---|---|---|---|---|
| Explanatory Variable | Yes<br>(N=xx) | No<br>(N=xx) | Odds-Ratio<br>[95% CI] | p-value | Odds-Ratio<br>[95% CI] | p-value |
| n | XX | XX | | | | |
| Missing data | Х | X | | | | |
| Factor 1 (qualitative) | | | | x.xxx | | x.xxx |
| Modality 1 (reference) | xx (xx.x%) | xx (xx.x%) | 1.00 | | 1.00 | |
| Modality 2 | xx (xx.x%) | xx (xx.x%) | x.xx [x.xx;x.xx] | | x.xx [x.xx;x.xx] | |
| Factor 2 (quantitative) | | | | X.XXX | | x.xxx |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | | | | |
| Per XX-unit increment | | | x.xx [x.xx;x.xx] | | x.xx[x.xx;x.xx] | |

#### 10 REFERENCES

NA

#### 11 APPENDICES

#### 11.1 APPENDIX 1: DATA DERIVATION DETAILS

Age = (Patient screening visit date – Birthdate + 1) /365.25, where day of birth is imputed to 15, as only month and year of birth are recorded.

Diastolic Blood Pressure classes:

- < 60 mmHg,
- [61 70] mmHg,
- [71 80] mmHg,
- [81 90] mmHg,
- [91 100] mmHg,
- > 100 mmHg.

#### Heart Rate classes:

- < 50 bpm,
- [51-60] bpm,
- [61 70] bpm,
- [71 80] bpm,
- [81 90] bpm,
- [91 100] bpm,
- [101 120] bpm,
- > 120 bpm.

#### PR interval classes:

- [90 100] ms
- [101 110] ms
- [111 120] ms
- [121 130] ms
- [131 140] ms
- [141 150] ms
- [151 160] ms
- [161 170] ms
- [171 180] ms
- [181 190] ms
- [191 200] ms
- [201 210] ms
- [211 220] ms
- [221 230] ms

- [231 240] ms
- [241 250] ms
- [251 260] ms
- [261 270] ms
- [271 280] ms
- > 280 ms

# Serum Free Light Chain Ratio:

sFLC Ratio = Kappa / Lambda,

# sFLC ratio classes:

- < 0.26,
- [0.26 1.65],
- > 1.65.

Abormal values for all quantitative variables will be defined after medical advise.